CLINICAL TRIAL: NCT03070977
Title: Interprofessional Training in a Psychiatric Study Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric Research Unit, Region Zealand, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Sidse Arnfred, Clinical Research Associate Professor in Psychiatry, MD MSc PhD DMSc Dep. Of Clinical Medicine, Faculty of Health and Medicine, University of Copenhagen and Psychiatric Department Slagelse, Region Zealand, Denmark., Psychiatric Research Unit, Region Zealand, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PRURegionZealand
Record Dates: First submitted 2017-01-21; First posted 2017-03-06 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Interdisciplinary Communication
Keywords: Interprofessional education; Training unit; Psychiatry; Patient reported outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interprofessional study unit (Experimental): In 2015, Psychiatry in Slagelse established an interprofessional clinical training unit. The aim was to create a new environment for learning, where students could learn from each other and develop competence in interprofessional collaboration. In the training unit there are more students than in the other standard psychiatric wards and several professions are included.
  Interventions: Other: Interprofessional clinical training unit
- Standard unit (No Intervention): Students in the control group receive training in standard psychiatric wards.

INTERVENTIONS:
Other: Interprofessional clinical training unit — In 2015, Psychiatry in Slagelse established an interprofessional clinical training unit. The aim was to create a new environment for learning, where students could learn from each other and develop competence in interprofessional collaboration. In the training unit there are more students than in the other standard psychiatric wards and several professions are included.
  A facilitator team is responsible for the interprofessional training. In autumn 2016 seven professionals participate in course of facilitating interprofessional collaboration and training. The intervention involved the total staff participation in an initial workshop.
  The training unit is based on two educational interventions: Student participation in clinical care teams and interprofessional group tuition sessions.
  Arms: Interprofessional study unit

SUMMARY:
Research question and basic idea:

Interprofessional collaboration is a skill that many health professionals need to develop. Interprofessional training offers a way to improve collaboration and patient care. The increasing number of psychiatric patients with complex needs, requires mental healthcare providers to enhance their skills. It necessitates that healthcare professionals collaborate effectively; nevertheless, many have not been trained in an interprofessional environment. Health professionals lack sufficient knowledge of other professional roles and competences to engage in teamwork. Interprofessional training units have been designed to create an optimal learning environment for healthcare students. These training units provide a new environment for learning, where students can learn from each other and develop competence in interprofessional collaboration. This collaboration gives students from several health professions an opportunity to achieve a greater understanding of the overall picture of the patient´s life. The limited data available suggest interprofessional collaboration interventions can improve health-care processes and outcomes; however, better designed studies are needed.

Objective: Therefore, we will investigate whether placement at a psychiatric training unit compared with placement at a standard psychiatric ward improves students' interprofessional skills and patients' health status and satisfaction.

DETAILED DESCRIPTION:
Research question and basic idea:

Interprofessional collaboration is a skill that many health professionals need to develop. Interprofessional training offers a way to improve collaboration and patient care. The increasing number of psychiatric patients with complex needs, requires mental healthcare providers to enhance their skills. It necessitates that healthcare professionals collaborate effectively; nevertheless, many have not been trained in an interprofessional environment. Health professionals lack sufficient knowledge of other professional roles and competences to engage in teamwork. Interprofessional study units have been designed to create an optimal learning environment for healthcare students. These study units provide a new environment for learning, where students can learn from each other and develop competence in interprofessional collaboration. This collaboration gives students from several health professions an opportunity to achieve a greater understanding of the overall picture of the patient´s life. The limited data available suggest interprofessional collaboration interventions can improve health-care processes and outcomes; however, better designed studies are needed.

Objective: Therefore, we will investigate whether placement at a psychiatric training unit compared with placement at a standard psychiatric ward improves students' interprofessional skills and patients' health status and satisfaction.

Methods Design We designed a non-randomized intervention study with an intervention group (interprofessional training unit) and a comparison group (conventional inpatient ward). Patients were included in the period October 2016 - March 2018. The two wards were comparable in terms patient categories (psychiatric diagnoses), and the size, staffing and design of wards (17 single-bed rooms in each ward). Students in the intervention group receive interprofessional training in the training unit in Slagelse (SL3), while students in the comparison group receive conventional training in a standard wards (SL2,SL4,SL5). The intervention is an interprofessional clinical training unit including students from nursing, medicine, psychology, social work and nursing assistants.

Questionnaires were administered to both groups at the beginning (T1) and end of hospitalization (T2).

Sample size and feasibility:

We powered the trial at 80% (α=0.05) to detect an effect size of 0.4, which we regarded as reasonable for determining clinically meaningful differences between interventions. Based on the power calculation we needed 120 patients per group Likewise, we conducted a power calculation regarding the students based on findings in a cross-sectional study. We used the students' interprofessional skills as the primary outcome. In the cross-sectional study the students had a mean score (RIPLS) of 69.98 (SD 25.5). When the sample size was calculated, 70 students were needed in both the intervention and the control group. 82 students have clinical placement in the psychiatric study unit in Slagelse annually (SL3) and 67 students have clinical placement in the standard psychiatric wards (SL2, SL4 and SL5). Therefore, it seems realistic to include 190 students within 18 months.

Participants:

Students taking part in their clinical placement in Psychiatry West in Slagelse. Primarily including students from Nursing, in their 3rd year clinical placement, graduate medical students 4th term, clinical placement in psychiatry and nursing assistants in their 2nd year clinical placement. Students from the intervention group are similar to the comparison group in terms of stage of education and duration of clinical training.

Inpatients aged 18-65 suffering from psychiatric disorders such as schizophrenia, psychosis, major depression, bipolar disorder, or severe personality disorder, and admitted October 2016 - March 2018, were included.

Allocation and recruitment:

After primary admission in the emergency ward, the patients were referred to inpatient wards based on their home address.

Students in both groups are allocated by program coordinators and supervisors from the involved university and colleges (University of Copenhagen, University College Zealand and Social and Healthcare College Zealand). The supervisors are responsible for the two groups of students and provided lists of names.

Data were entered into the EasyTrial © online Clinical Trial Management system. Data were labelled with unique identifiers, and all personal identifiers were removed or disguised during analysis to preclude personal identification.

Intervention:

In 2015, Psychiatry in Slagelse established an interprofessional clinical training unit. The aim was to create a new environment for learning, where students could learn from each other and develop competence in interprofessional collaboration. In the training unit there are more students than in the other standard psychiatric wards and several professions are included.

A facilitator team is responsible for the interprofessional training. In autumn 2016 seven professionals participate in course of facilitating interprofessional collaboration and training. The intervention involved the total staff participation in an initial eight-hour interactive workshop on the subject.

The training unit is based on two educational interventions: Student participation in clinical care teams and interprofessional group tuition sessions.

Clinical care team:

The interprofessional clinical care team ensures that the patient pathways are well-planned and well-coordinated. Professionals included in the patient's care are part of the team alongside with the patient and their relatives. In the training unit the students are also part of the team. The team meets weekly. The team conference is an important interdisciplinary element in support of patient care during hospitalization. This is very important as patients' needs are often complex.

Interprofessional group tuition:

Interprofessional group tuition is a method to improve professional reflection on clinical practice. Patients in the training unit and their treatment and care are in focus. The group tuition takes an entire day with a mixture of theory and patient cases, in which all professional groups of students participate. The supervisors are responsible for planning the sessions.

Ethical considerations:

The study is licensed by the Danish Data Protection Agency (2008-58-0020) and needed no further ethical approval according to Danish legislation (16-000014). Data is anonymized and stored in a secure server. Students and patients will be informed about the project and its purpose immediately before participation. The return of questionnaires will be considered consent to participation.

Time schedule:

Data collection is started October 2016 and will run for 18 months. Data analysis will start January 2018. Publications are planned for 2018. The PhD study is scheduled for 3 years and will end on 31 March 2019.

ELIGIBILITY:
Inclusion Criteria:

* Students: Health care students in clinical practice from November 2016 - 30 April 2018.
* Patients: Inpatients aged 18-65 suffering from psychiatric disorders such as schizophrenia, psychosis, major depression, bipolar disorder, or severe personality disorder, and admitted October 2016 - March 2018, were included.

Exclusion Criteria:

* Patients: Patients, who did not consent to participation or failed to complete the questionnaire at the beginning of their stay, were excluded from the study. In addition, patients hospitalized for less than a week, were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
The effect on students' interprofessional skills. | Week 9-10 after placement onset
  We use the Readiness for Inter Professional Learning Scale (RIPLS): The 29 item questionnaire has four subscales assessing; Teamwork and Collaboration, Negative Professional Identity, Positive Professional Identity, and Roles and Responsibilities.
  Score range from 29 to 145, with higher scores indicating higer level of readiness of interprofessional learning.
Health status | Three weeks after admission
  We use Short Form Health Survey (SF-36) to assess the patients' self-reported health status. On the basis of the questionnaire's 36 items, we calculated two summary scores; the physical component score and the mental component score (PCS and MCS, respectively). Scores range from 0 (zero) to 100, with higher scores indicating better health.
Psychological distress | Three weeks after admission
  We use The Kessler Psychological Distress Scale (K10). Its 10 items measure the experienced level of anxiety and depressive symptoms over the preceding four weeks, with a score range from 10 to 50, higher scores indicating more anxiety and stronger depressive symptoms.

SECONDARY OUTCOMES:
The effect on students' interprofessional team collaboration Scale | Week 9-10 after placement onset
  We use the Assessment of Interprofessional Team Collaboration Scale (AITCS): Including 37 items distributed on 3 subscales; Partnership/Shared decision making, Cooperation, and Coordination. With a score range from 37 to 185, higher scores indicating higher level of collaboration.
Patient Satisfaction | Three weeks after admission
  We use the Client Satisfaction Questionnaire, 8 item version (CSQ-8). Total scores range from 8 to 32, with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Sidse Arnfred, MD, Dr.med, Principal Investigator — Psychiatric Research Unit, Region Zealand, Denmark
Locations (1):
- Psychiatry in Slagelse, Slagelse, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reeves S. A systematic review of the effects of interprofessional education on staff involved in the care of adults with mental health problems. J Psychiatr Ment Health Nurs. 2001 Dec;8(6):533-42. doi: 10.1046/j.1351-0126.2001.00420.x. PMID 11842481
- [Background] Pauze E, Reeves S. Examining the effects of interprofessional education on mental health providers: Findings from an updated systematic review. J Ment Health. 2010 Jun;19(3):258-71. doi: 10.3109/09638230903469244. PMID 20441490
- [Background] Reeves S, Perrier L, Goldman J, Freeth D, Zwarenstein M. Interprofessional education: effects on professional practice and healthcare outcomes (update). Cochrane Database Syst Rev. 2013 Mar 28;2013(3):CD002213. doi: 10.1002/14651858.CD002213.pub3. PMID 23543515
- [Background] Zwarenstein M, Bryant W. Interventions to promote collaboration between nurses and doctors. Cochrane Database Syst Rev. 2000;(2):CD000072. doi: 10.1002/14651858.CD000072. PMID 10796485
- [Background] Reeves S, Zwarenstein M, Goldman J, Barr H, Freeth D, Hammick M, Koppel I. Interprofessional education: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD002213. doi: 10.1002/14651858.CD002213.pub2. PMID 18254002
- [Background] Hammick M, Freeth D, Koppel I, Reeves S, Barr H. A best evidence systematic review of interprofessional education: BEME Guide no. 9. Med Teach. 2007 Oct;29(8):735-51. doi: 10.1080/01421590701682576. PMID 18236271
- [Background] Young AS, Chinman M, Forquer SL, Knight EL, Vogel H, Miller A, Rowe M, Mintz J. Use of a consumer-led intervention to improve provider competencies. Psychiatr Serv. 2005 Aug;56(8):967-75. doi: 10.1176/appi.ps.56.8.967. PMID 16088014
- [Background] Priest HM, Roberts P, Dent H, Blincoe C, Lawton D, Armstrong C. Interprofessional education and working in mental health: in search of the evidence base. J Nurs Manag. 2008 May;16(4):474-85. doi: 10.1111/j.1365-2834.2008.00867.x. PMID 18405264
- [Background] Ponzer S, Hylin U, Kusoffsky A, Lauffs M, Lonka K, Mattiasson AC, Nordstrom G. Interprofessional training in the context of clinical practice: goals and students' perceptions on clinical education wards. Med Educ. 2004 Jul;38(7):727-36. doi: 10.1111/j.1365-2929.2004.01848.x. PMID 15200397
- [Background] Reeves S, Freeth D, McCrorie P, Perry D. 'It teaches you what to expect in future . . . ': interprofessional learning on a training ward for medical, nursing, occupational therapy and physiotherapy students. Med Educ. 2002 Apr;36(4):337-44. doi: 10.1046/j.1365-2923.2002.01169.x. PMID 11940174
- [Background] Jacobsen F, Fink AM, Marcussen V, Larsen K, Hansen TB. Interprofessional undergraduate clinical learning: results from a three year project in a Danish Interprofessional Training Unit. J Interprof Care. 2009 Jan;23(1):30-40. doi: 10.1080/13561820802490909. PMID 19142781
- [Background] Hylin U, Nyholm H, Mattiasson AC, Ponzer S. Interprofessional training in clinical practice on a training ward for healthcare students: a two-year follow-up. J Interprof Care. 2007 Jun;21(3):277-88. doi: 10.1080/13561820601095800. PMID 17487706
- [Background] Coster S, Norman I, Murrells T, Kitchen S, Meerabeau E, Sooboodoo E, d'Avray L. Interprofessional attitudes amongst undergraduate students in the health professions: a longitudinal questionnaire survey. Int J Nurs Stud. 2008 Nov;45(11):1667-81. doi: 10.1016/j.ijnurstu.2008.02.008. Epub 2008 Apr 18. PMID 18423644
- [Derived] Marcussen M, Norgaard B, Borgnakke K, Arnfred S. Improved patient-reported outcomes after interprofessional training in mental health: a nonrandomized intervention study. BMC Psychiatry. 2020 May 14;20(1):236. doi: 10.1186/s12888-020-02616-x. PMID 32410668
- [Derived] Marcussen M, Norgaard B, Borgnakke K, Arnfred S. Interprofessional clinical training in mental health improves students' readiness for interprofessional collaboration: a non-randomized intervention study. BMC Med Educ. 2019 Jan 18;19(1):27. doi: 10.1186/s12909-019-1465-6. PMID 30658648